CLINICAL TRIAL: NCT05332795
Title: The Impact of Metformin on the Outcome of Gouty Arthritis in a Cohort of Egyptian Gouty Patients.
Acronym: Mets in gout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Dalia Salah Saif, Assistant professor of physical medicine,rheumatology and rehabilitation., Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1478
Record Dates: First submitted 2022-04-02; First posted 2022-04-18 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Gouty Arthritis
MeSH Terms: conditions — Arthritis, Gouty | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1: gouty patients on metformin. (Active Comparator): metformin users: include gouty patients, who will receive metformin tablets (1000 mg) once daily for about 3 months.
  Interventions: Drug: Metformin
- gouty patients on placebo. (Placebo Comparator): placebo users: include gouty patients, who were on placebo tablets once daily for about 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — gouty patients, will receive metformin tablets (1000 mg) once daily for about 3 months.
  Arms: group 1: gouty patients on metformin.
Drug: Placebo — gouty patients, will receive placebo tablets once daily for about 3 months.
  Arms: gouty patients on placebo.

SUMMARY:
Objective:

To study the impact of metformin on the outcome of gouty arthritis in a cohort of Egyptian gouty patients, and to evaluate its effect on local joint inflammation, inflammatory cytokines (IL-1β and IL-6), and life quality.

Methods:

A prospective randomized, single-blinded parallel randomized control study included 100 patients with active inflammatory gouty arthritis were randomized to receive metformin (1000mg/day) or placebo in addition to the traditional lines of treatment of gout. The clinical and laboratory data of the patients will be analyze at baseline, then after 3, and 6 months, with the assessment of gout disease activity, in addition, serum IL-1β and IL-6, the number of attacks per year, treatment satisfaction, quality of life, and disability index were evaluated at the 6th month from starting metformin and placebo therapy.

DETAILED DESCRIPTION:
Background: Metformin has anti-inflammatory properties, as it suppresses the inflammatory process by down-regulating the transcription factor, nuclear factor kappa B (NF-kB), through AMP-activated protein kinase (AMPK)-dependent and independent pathways.

Objective:

To study the impact of metformin on the outcome of gouty arthritis in a cohort of Egyptian gouty patients, and to evaluate its effect on local joint inflammation, inflammatory cytokines (IL-1β and IL-6), and life quality.

Methods:

A prospective randomized, single-blinded parallel randomized control study included 100 patients with active inflammatory gouty arthritis were randomized to receive metformin (1000mg/day) or placebo in addition to the traditional lines of treatment of gout. The clinical and laboratory data of the patients will be analyzed at baseline, then after 3, and 6 months, with the assessment of gout disease activity, in addition, serum IL-1β and IL-6, the number of attacks per year, treatment satisfaction, quality of life, and disability index were evaluated at the 6th month from starting metformin and placebo therapy.

ELIGIBILITY:
Inclusion Criteria:

* gouty patients who fulfilled the American College of Rheumatology clinical criteria.
* gouty patients with active inflammatory arthritis.

Exclusion Criteria:

* Patients with any type of inflammatory arthritis.
* Patients with systemic disease as diabetes, hypertension,
* Patients with hyperlipidemia, coronary artery disease,
* Patients with renal or hepatic insults,
* pregnant and lactating females

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Serological remission criteria | at 3 months post intervention.
  by measuring serum uric acid for patients of the present study, it must be less than 6 mg/dL.
Articular remission criteria | at 3 months post intervention.
  by examining the number of swollen and tender joints score, they must be less than 2 tender and swollen joints..
Clinical remission criteria | at 3 months post intervention.
  by assessing the grade of joint pain, it must be reduced from the first visit(regarding Visual analogue scale

SECONDARY OUTCOMES:
Gout Impact Scale (GIS) | at 3 months post intervention.
  by measuring GIS score, as higher scores in the GIS (range 0-100) imply a greater restriction of activity and a greater impact of gout and vice versa.

OTHER OUTCOMES:
Health-related quality of life HRQOL | at 3 months post intervention.
  Health-related quality of life HRQOL was assessed using the SF-36 subscale of physical functioning (PF-10), as Lower PF-10 scores (range 0-100) imply more functional limitations, and vice versa.

CONTACTS AND LOCATIONS:
Locations (1):
- Dalia Salah Saif, Menoufia Governorate, MD, Egypt

IPD SHARING:
Plan to Share IPD: Undecided